CLINICAL TRIAL: NCT04340063
Title: Amplify Gait to Improve Locomotor Engagement in Spinal Cord Injury (AGILE SCI) Trial
Brief Title: Amplify Gait to Improve Locomotor Engagement in Spinal Cord Injury
Acronym: AGILE SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B3371-R; I01RX003371 (NIH)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: gait; locomotion; walking; balance; spinal cord injury; rehabilitation robotics
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a two-arm parallel assignment intervention. Participants will be randomized into a high intensity locomotor training intervention that will be conducted in either a normal treadmill environment or in a movement amplification environment.
Who Masked: Outcomes Assessor
Masking Description: Study personnel performing the clinical assessments will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treadmill group (Active Comparator): Participants randomized to the Treadmill group will complete high intensity gait training on a treadmill.
  Interventions: Device: Gait training performed on a treadmill
- Movement Amplification group (Experimental): The locomotor training protocol described for the Treadmill group will be used for the Movement Amplification group with one exception. The Movement Amplification group will perform all gait training within the movement amplification environment.
  Interventions: Device: Gait training performed in a Movement Amplification Environment

INTERVENTIONS:
Device: Gait training performed on a treadmill — Participants randomized to the Control group will complete high intensity gait training on a treadmill.
  Other Names: Treadmill Group
  Arms: Treadmill group
Device: Gait training performed in a Movement Amplification Environment — The Experimental group will perform all gait training within the movement amplification environment. To create the movement amplification environment, the investigators have constructed a cable-driven robot, the Agility Trainer. The Agility Trainer applies small forces to the pelvis that increase the difficulty to maintain forward walking
  Other Names: Movement Amplification Group
  Arms: Movement Amplification group

SUMMARY:
Spinal cord injury (SCI) affects ~42,000 Veterans. The VA provides the single largest network of SCI care in the nation. The lifetime financial burden of SCI can exceed $3 million. A major cost of SCI is impaired mobility. Limited mobility contributes to decreased ability to work, increased care requirements, secondary injury, depression, bone mineral density loss, diabetes, and decreased cardiovascular health. Among ambulatory individuals with iSCI, residual balance deficits are common and are strongly correlated with both functional walking ability and participation in walking activities. The development of effective rehabilitation tools to improve dynamic balance would substantially improve quality of life for Veterans living with iSCI. Improving mobility through interventions that enhance dynamic balance would positively impact health, independence, and the ability to integrate into social, intellectual, and occupational environments.

DETAILED DESCRIPTION:
Background:

Among ambulatory individuals with incomplete spinal cord injury (iSCI), residual balance deficits are common and are a primary factor limiting participation in walking activities. There is broad recognition that effective evidence-based interventions are needed to enhance dynamic balance following iSCI. However, improving dynamic balance after iSCI has proven to be very challenging. Experimental interventions that amplify self-generated movements (e.g. error augmentation) may accelerate motor learning by intensifying sensory motor feedback and facilitating exploration of alternative motor control strategies. These features may be beneficial for retraining dynamic balance after iSCI. The investigators have developed a cable-driven robot to create a movement amplification environment during treadmill walking by applying a continuous viscous force field to the pelvis that is proportional in magnitude to a participant's real-time range of motion (ROM) velocity. The purpose is to investigate if locomotor training performed in a movement amplification environment can effectively improve dynamic balance and increase participation in walking activities of individuals with iSCI.

Specific Aims:

Aim 1: To evaluate if locomotor training performed in a movement amplification environment is effective for improving dynamic balance of individuals with iSCI. The investigators' pilot data found that following locomotor training performed in a movement amplification environment three individuals with iSCI each improved dynamic balance by more than 30%. These improvements were accompanied by faster over ground walking speeds and improved reactive balance. Thus, the investigators hypothesize that improvements in dynamic balance during walking will be greater when locomotor training is performed in a movement amplification environment when compared to locomotor training performed in a traditional treadmill environment.

Aim 2: To evaluate the impact of locomotor training performed in either a movement amplification environment or in a traditional treadmill environment on participation in walking activities. Based on evidence identifying a strong relationship between balance and steps per day in ambulatory individuals with iSCI, the investigators hypothesize that training in the movement amplification environment will positively impact dynamic balance, and in turn increase participating in walking activities.

Approach:

The investigators will conduct a two-arm parallel-assignment intervention and will enroll 36 ambulatory participants with chronic motor incomplete spinal cord injury. Participants will be randomized into either a Control group receiving locomotor training or an Experimental group receiving locomotor training performed in a movement amplification environment. All participants will receive 20 training sessions. The investigators will assess changes in dynamic balance using measures that span the International Classification of Functioning, Disability and Health (ICF) framework including; 1) clinical outcome measures of gait, balance, and quality of life, 2) biomechanical assessments of the capacity to control center of mass (COM) motion during walking, and 3) data collected from activity monitors to quantify changes in participation in walking activities as evaluated by number of steps taken per day.

Impact:

Training dynamic balance of individuals with iSCI by amplifying their own self-generated center of mass motion during walking is a radical departure from current practice and may create effective new clinical strategies for addressing balance impairments of individuals with iSCI. Successful outcomes from the proposed trial would motivate development of clinically-feasible tools to first replicate and then to evaluate the movement amplification environment within the VA's clinical care settings. Knowledge gained from this study will expand the understanding of how individuals with iSCI learn dynamic balance and how targeted dynamic balance training impacts participation in walking activities.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable with medical clearance from a physician to participate
* Neurologic level of the SCI between C1-T10 with American Spinal Injury Association (ASIA) Impairment Scale (AIS) C or D
* > 6 months since initial injury
* Passive range of motion of the legs within functional limits and not restricting the ability to engage in locomotor training
* Able to ambulatory 10m with no physical assistance, use of assistive devices (e.g. single cane, rolling walker), and/or braces that do not cross the knee joint (e.g. ankle foot orthosis) are permitted
* Able to provide transportation to and from the testing location.

Exclusion Criteria:

* Excessive spasticity in the lower limbs as measured by a score of > 3 on the Modified Ashworth Scale
* Inability to tolerate 30 minutes of standing
* Severe cardiovascular and pulmonary disease
* History of recurrent fractures or known orthopedic problems in the lower extremities (i.e. heterotopic ossification)
* Concomitant central or peripheral neurological injury (i.e. traumatic head injury or peripheral nerve damage in lower limbs)
* Inability to provide informed consent due to cognitive impairments
* Presence of unhealed decubiti or other skin compromise
* Enrollment in concurrent physical therapy or research involving locomotor training
* Use of braces/orthotics crossing the knee joint
* Known pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith E Gordon, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will create and share de-identified, anonymized data sets. Data sets will be open file formats that include documentation of the material. The investigators will link data sets to associated study publications. Final data sets will be made available as per Hines VA Hospital local policy for long term storage and access until enterprise-level resources become available. These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.
  The final data sets will be sufficient for anyone to perform analogous or supplemental analyses that would permit validation of the analysis and results.
  The sharing of data will enable others to evaluate the data and to validate and interpret the data independently.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following the completion and publication of study results.
Access Criteria: Data will be publicly available.

REFERENCES:
- [Derived] Gordon KE, Dusane S, Kahn JH, Shafer A, Brazg G, Henderson H, Kim KA. Amplify Gait to Improve Locomotor Engagement in Spinal Cord Injury (AGILE SCI) trial: study protocol for an assessor blinded randomized controlled trial. BMC Neurol. 2024 Aug 3;24(1):271. doi: 10.1186/s12883-024-03757-2. PMID 39097695

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 participants signed the consent form. Out of 38, 2 participants were excluded as they did not meet the inclusion criteria at in person screening and were not assigned to any group.
Groups:
- Treadmill Group: Participants randomized to the Treadmill group will complete high intensity gait training on a treadmill in a natural environment without forces applied (control group).
- Movement Amplification Group: The locomotor training protocol described for the Treadmill group will be used for the Movement Amplification group with one exception. The Movement Amplification group will perform all gait training within the movement amplification environment.
  The Experimental group will perform all gait training within the movement amplification environment. To create the movement amplification environment, the investigators have constructed a cable-driven robot, the Agility Trainer. The Agility Trainer applies small forces to the pelvis that increase the difficulty to maintain forward walking
Period: Overall Study
Arm/Group | Treadmill Group | Movement Amplification Group
Started | 18 | 18
Pre-training Assessment | 18 | 18
Mid-training Assessment | 14 | 16
Post-training Assessment | 14 | 16
Follow-up Assessment | 14 | 14
Completed | 14 | 14
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treadmill Group High Initial Function: Participants randomized to the Treadmill group will complete high intensity gait training on a treadmill in a natural environment without any forces applied (control group).
- Movement Amplification Group High Initial Function: The locomotor training protocol described for the Treadmill group and stratified into high initial function (who walk ≥0.5m/s without the use of any assistive device) will be used for the Movement Amplification group with one exception. The Movement Amplification group will perform all gait training within the movement amplification environment.
  Gait training performed in a Movement Amplification Environment: The Experimental group will perform all gait training within the movement amplification environment. To create the movement amplification environment, the investigators have constructed a cable-driven robot, the Agility Trainer. The Agility Trainer applies small forces to the pelvis that increase the difficulty to maintain forward walking
- Total: Total of all reporting groups
Arm/Group | Treadmill Group High Initial Function | Movement Amplification Group High Initial Function | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.44 (19.79) | 54.61 (17.52) | 54.03 (18.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 15 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 11 | 16 | 27
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 10 | 11 | 21
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 0 | 2
Time Since Injury [Mean (Standard Deviation); unit: years] | 10.56 (14.96) | 7.94 (8.83) | 9.25 (12.18)

OUTCOME MEASURES:

1. Primary Outcome: Functional Gait Assessment (FGA)
Description: The FGA is a ten-item test that evaluates dynamic balance and postural stability during gait. Each item on the test is scored from 0 (severe impairment) to 3 (normal ambulation). Total score of this test is 30, with higher score indicating better walking balance. Lowest possible score is 0.
Time Frame: Pre-training assessment (Baseline), Mid-training assessment (after 10 sessions, ~5 weeks from Baseline), Post-training assessment (after 20 sessions, ~10 weeks from Baseline), Follow-up assessment (3 month from Post, ~6 months from Baseline)
Population: A total of 36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 15.22 (7.82) | 14.22 (7.61)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 19.38 (7.31) | 18.13 (7.16)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 20.29 (7.94) | 19.88 (7.64)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 20.57 (8.08) | 21.00 (7.87)
Statistical Analysis 1: Comparison: Treadmill Group vs Movement Amplification Group; A linear mixed-effects model (LMM) evaluated the effect of training (pre-, mid-, and post- assessments). Random effect of participant was used and fixed effects were time (assessment order) and a time by group interaction (Treadmill or Movement Amplification). A binomial distribution was used for this model; Test type: Other; p < 0.001, Mixed Models Analysis — Effect of time (pre-, mid-, and post- assessments); Odds Ratio, log = 0.4, 95% CI 2-sided [0.25 to 0.55]
Statistical Analysis 2: Comparison: Treadmill Group vs Movement Amplification Group; Test type: Other; p = 0.8, Mixed Models Analysis — Interaction effect for time (pre-, mid-, and post- assessments) by group (Movement Amplification); Odds Ratio, log = -0.03, 95% CI 2-sided [-0.22 to 0.16]
Statistical Analysis 3: Comparison: Treadmill Group vs Movement Amplification Group; A linear mixed-effects model (LMM) evaluated the post-training and follow-up assessments if an effect was found during training. Random effect of participant and fixed effects of time (assessment order) and the time by group (Treadmill or Movement Amplification) interaction were used. A binomial distribution was used for this model; Test type: Other; p = 0.5, Mixed Models Analysis — Effect of time (post-training and follow-up assessments); Odds Ratio, log = 0.09, 95% CI 2-sided [-0.18 to 0.36]
Statistical Analysis 4: Comparison: Treadmill Group vs Movement Amplification Group; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.6, Mixed Models Analysis — Interaction effect of time (post-training and follow-up assessments) by group (Movement Amplification); Odds Ratio, log = -0.07, 95% CI 2-sided [-0.31 to 0.17]

2. Primary Outcome: Lateral Center of Mass Excursion
Description: The investigators will perform biomechanical laboratory assessments to make quantitative measures of changes in dynamic balance during walking. The investigators will record 3D coordinates of reflective markers placed on anatomical landmarks. These markers will be used to quantify changes in an individual's average lateral center of mass excursion occurring each stride during treadmill walking.
Time Frame: as for outcome 1
Population: A total of 35 participants were analyzed
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 17
centimeters
  Pre-training assessment | 10.16 (4.5) | 9.82 (3.68)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 8.51 (3.75) | 7.42 (2.39)
  Post-training assessment: number analyzed (Participants) | 14 | 15
  Post-training assessment | 8.43 (4.35) | 7.19 (2.23)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 8.73 (4.2) | 7.38 (1.73)
Statistical Analysis 1: Comparison: Treadmill Group vs Movement Amplification Group; A linear mixed-effects model (LMM) evaluated the effect of training (pre-, mid-, and post- assessments). Random effect of participant and fixed effects of time (assessment order) and time by group (Treadmill or Movement Amplification) interaction were used; Test type: Other; p = 0.8, Mixed Models Analysis — Effect of time (pre-, mid-, and post- assessments); Slope = 0.06, 95% CI 2-sided [-0.50 to 0.62]
Statistical Analysis 2: Comparison: Treadmill Group vs Movement Amplification Group; A linear mixed-effects model (LMM) evaluated the effect of training (pre-, mid-, and post- assessments). Random effect of participant and fixed effects of time (assessment order) and the time by group (Treadmill or Movement Amplification) interaction were used; Test type: Other; p = 0.012, Mixed Models Analysis — Interaction effect of time by group (Movement Amplification); Slope = -0.7, 95% CI 2-sided [-1.2 to -0.16]
Statistical Analysis 3: Comparison: Treadmill Group vs Movement Amplification Group; A linear mixed-effects model (LMM) evaluated the post-training and follow-up assessments if an effect was found during training. Random effect of participant and fixed effects of time (assessment order) and the time by group (Treadmill or Movement Amplification) interaction were used; Test type: Other; p = 0.3, Mixed Models Analysis — Effect of time (post-training to follow-up); Slope = 0.26, 95% CI 2-sided [-0.22 to 0.75]
Statistical Analysis 4: Comparison: Treadmill Group vs Movement Amplification Group; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.4, Mixed Models Analysis — Interaction effect of time (post-training to follow-up) by group; Slope = -0.20, 95% CI 2-sided [-0.69 to 0.29]

3. Primary Outcome: Daily Stepping
Description: The investigators will assess the amount of daily stepping in the home and community during three 1-week periods. Daily stepping will be measured and recorded using an activity monitor. HIgher number of daily stepping indicates greater physical activity levels or greater walking in the community setting.
Time Frame: Pre-training assessment (Baseline), Post-training assessment (after 20 sessions, ~10 weeks from Baseline), Follow-up assessment (3 month from Post, ~6 months from Baseline)
Population: A total of 36 participants were analyzed. 1 participant's data not collected at Baseline but included in later assessment periods.
Measure: Mean (Standard Deviation); unit: Average steps per day
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
Average steps per day
  Pre-training assessment: number analyzed (Participants) | 17 | 18
  Pre-training assessment | 5,680 (4,945) | 3,264 (3,081)
  Post-training assessment: number analyzed (Participants) | 13 | 16
  Post-training assessment | 5,480 (4,792) | 4,284 (3,039)
  Follow-up assessment: number analyzed (Participants) | 14 | 13
  Follow-up assessment | 6,041 (4,421) | 3,530 (2,524)
Statistical Analysis 1: Comparison: Treadmill Group vs Movement Amplification Group; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.9, Mixed Models Analysis — Effect of time (pre-, mid-, and post- assessments); Slope = -52, 95% CI 2-sided [-651 to 456]
Statistical Analysis 2: Comparison: Treadmill Group vs Movement Amplification Group; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.8, Mixed Models Analysis — Interaction effect of time by group (Movement Amplification); Slope = 79, 95% CI 2-sided [-622 to 780]

4. Secondary Outcome: 10 Meter Walk Test (10MWT)_Fast Speed
Description: The 10MWT is a simple measurement of an individuals average walking speed.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: meter per second
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
meter per second
  Pre-training assessment | 0.86 (0.51) | 0.87 (0.52)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 1.14 (0.68) | 1.01 (0.53)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 1.15 (0.61) | 1.08 (0.48)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 1.16 (0.64) | 1.09 (0.51)

5. Secondary Outcome: 10 Meter Walk Test (10MWT)_Preferred Speed
Description: The 10MWT is a simple measurement of an individuals average walking speed.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: meter per second
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
meter per second
  Pre-training assessment | 0.65 (0.40) | 0.65 (0.38)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 0.83 (0.45) | 0.72 (0.38)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 0.83 (0.41) | 0.79 (0.35)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 0.84 (0.41) | 0.81 (0.37)

6. Secondary Outcome: Activities Specific Balance Confidence (ABC) Scale
Description: The ABC scale is a 16-item self-report measurement of an individual's confidence while performing numerous postural and ambulatory activities. Each item is rated on a scale of 0 (no confidence) to 100 (complete confidence). Overall score is calculated by adding item scores and then dividing by the total number of items. Total score is 100. Higher score indicates greater balance confidence i.e. ability to perform tasks with less or no fear of falling. Lowest possible score is 0.
Time Frame: as for outcome 1
Population: At post-training assessment, a total of 30 participants analyzed corresponds to those who completed intervention and post-training assessment. At follow up, a total of 28 participants analyzed corresponds to the participants who completed the intervention and follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 62.62 (22.96) | 65.39 (21.14)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 71.97 (22.94) | 75 (16.32)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 73.50 (25.46) | 74.06 (16.82)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 75.46 (24.77) | 77.32 (15.89)

7. Secondary Outcome: Balance Evaluations Systems Test (BESTest)
Description: The BESTest is used to assess balance impairments across six different domains of postural control. We will use only the reactive balance item from the BESTest to assess changes in the capacity to react to fore-aft, and lateral perturbations. Each item will be scored on a range from 0 (severe impairment) to 3 (no impairment). Highest score is 6 and lowest possible score is 0. Higher score indicates better ability to restore balance and better reactive stepping response during standing perturbation.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
units on a scale
  Pre-training assessment | 2.64 (1.98) | 1.88 (1.71)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 2.92 (2.14) | 2.13 (1.93)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 2.79 (2.42) | 2.40 (2.23)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 3.14 (2.35) | 2.71 (2.27)

8. Secondary Outcome: Berg Balance Scale (BBS)
Description: The BBS is a 14-item measure that assesses static balance. Each item is scored on a range of 0 to 4. A total score is determined by summing scores on the all the individual items. Total score is 56. Higher score indicates better static balance. Lowest possible score is 0.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 41.78 (11.95) | 41.67 (13.78)
  Mid-training assessment: number analyzed (Participants) | 13 | 16
  Mid-training assessment | 45.46 (11.09) | 46.63 (9.96)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 46.79 (9.68) | 48.38 (8.76)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 47.43 (9.21) | 48.64 (8.98)

9. Secondary Outcome: International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF)
Description: The ICIQ-UI SF is a 4-item self-report of urinary incontinence to document changes in bladder function. Scores range from 0-21, with greater values indicating increased severity.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 4.43 (5.2) | 4.19 (5.36)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 3.21 (4.51) | 3.63 (4.6)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 4.07 (5.08) | 4.31 (5.31)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 3.71 (4.7) | 4.57 (5.43)

10. Secondary Outcome: Lower Extremity Motor Score
Description: The lower extremity motor score assess strength of five muscle groups representing neurological levels L2 to S1. Muscle function is grade on a range from 0 (total paralysis) to 5 (active movement, full range of motion (ROM) against gravity and sufficient resistance to be considered normal. Total score is 50. Higher score indicates better or more complete motor function in the lower extremities. Lowest possible score is 0.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 39.33 (7.90) | 40.39 (6.06)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 41.14 (7.23) | 40.88 (6.24)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 41.71 (7.22) | 41.44 (6.16)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 42 (7.14) | 42 (5.91)

11. Secondary Outcome: Timed Up and Go (TUG)
Description: The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk. The participant sits in a chair with his/her back against the chair back. On the command "go," the patient rises from the chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down. Time to complete the task is reported. Participant must use the same assistive device each time he/she is tested to be able to compare scores.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
seconds
  Pre-training assessment: number analyzed (Participants) | 18 | 17
  Pre-training assessment | 34.18 (41.94) | 33.92 (39.28)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 21.49 (24.4) | 27.51 (32.55)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 23.59 (35.11) | 25.85 (36.82)
  Follow-up assessment: number analyzed (Participants) | 14 | 13
  Follow-up assessment | 21.24 (28.99) | 24.67 (28.59)

12. Secondary Outcome: Walking Index for Spinal Cord Injury II (WISCI II)
Description: The WISCI II evaluates the amount of physical assistance needed for gait after spinal cord injury. The index ranges from 0 (client is unable to stand and/or participate in assisted walking) to 20 (ambulates with no devices, no braces and no physical assistance, 10 meters). Highest score is 20 and lowest possible score is 0. Higher score indicates better ability to ambulate at least a distance of 10 meters without assistance from assistive device and/or from other person.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 16.17 (3.82) | 14.89 (4.65)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 17.57 (2.44) | 16.25 (3.86)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 18.00 (2.29) | 16.94 (3.79)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 18.21 (2.01) | 17.21 (4.10)

13. Secondary Outcome: The World Health Organization Quality of Life Scale (WHOQOL-BREF)_Physical
Description: The WHOQOL-BREF is a 26 item self-report quality of life assessment focusing on 4 different domains: physical, psychological, social relations and environment. The physical domain focuses on patients perception about his physical health including items related to mobility, daily activities, functional capacity, energy, pain, and sleep. Scores range from 0-100 with 100 indicating higher quality of life. Lowest possible score is 0.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 74.29 (18.56) | 62.63 (18.44)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 71.57 (17.66) | 55.69 (21.26)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 73.79 (14.25) | 65.06 (23.31)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 73.79 (20.02) | 59.57 (21.01)

14. Secondary Outcome: The World Health Organization Quality of Life Scale (WHOQOL-BREF)_Psychological
Description: The WHOQOL-BREF is a 26 item self-report quality of life assessment focusing on 4 different domains: physical, psychological, social relations and environment. The psychological domain focuses on patients perception about their psychological well-being, encompassing aspects like self-image, negative and positive feelings, self-esteem, and mental status. Scores range from 0-100 with 100 indicating higher quality of life. Lowest possible score is 0.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 76.00 (18.42) | 66.50 (16.94)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 75.93 (12.87) | 64.19 (22.81)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 78.07 (10.62) | 70.81 (22.26)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 76.79 (14.56) | 65.64 (20.87)

15. Secondary Outcome: The World Health Organization Quality of Life Scale (WHOQOL-BREF)_Social Relations
Description: The WHOQOL-BREF is a 26 item self-report quality of life assessment focusing on 4 different domains: physical, psychological, social relations and environment. The social relations domain focuses on patients perception about their social connections, support, and sexual life, contributing to their overall quality of life. Scores range from 0-100 with 100 indicating higher quality of life. Lowest possible score is 0.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 69.21 (21.18) | 60.56 (25.28)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 66.07 (18.70) | 62.94 (20.61)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 65.46 (17.47) | 57.81 (25.41)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 71.43 (18.48) | 59.79 (19.46)

16. Secondary Outcome: The World Health Organization Quality of Life Scale (WHOQOL-BREF)_Environment
Description: The WHOQOL-BREF is a 26 item self-report quality of life assessment focusing on 4 different domains: physical, psychological, social relations and environment. The environment domain focuses on patients perception about their surroundings, including factors like financial resources, safety, access to services, home environment, and the physical environment. social connections, support, and sexual life, contributing to their overall quality of life. Scores range from 0-100 with 100 indicating higher quality of life. Lowest possible score is 0.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Pre-training assessment | 80.50 (19.40) | 79.44 (16.65)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 77.86 (19.10) | 75.63 (20.44)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 80.93 (18.95) | 77.06 (19.72)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 84.00 (16.82) | 73.36 (19.13)

17. Secondary Outcome: Minimum Lateral Margin of Stability
Description: The investigators will perform biomechanical laboratory assessments to make quantitative measures of changes in dynamic balance during walking. The investigators will record 3D coordinates of reflective markers placed on anatomical landmarks. These markers will be used to quantify changes in an individual's average minimum lateral margin of stability (distance between a velocity weighted whole body center of mass position and the edge of the base of support) occurring each step during treadmill walking.
Time Frame: as for outcome 1
Population: A total of 35 participants were analyzed
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 17
centimeters
  Pre-training assessment | 5.84 (2.78) | 4.96 (2.4)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 6.16 (2.15) | 5.0 (3.23)
  Post-training assessment: number analyzed (Participants) | 14 | 15
  Post-training assessment | 6.33 (2.39) | 4.73 (3.48)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 6.32 (2.94) | 5.39 (3.42)

18. Secondary Outcome: Peak Lateral Center of Mass Speed
Description: The investigators will perform biomechanical laboratory assessments to make quantitative measures of changes in dynamic balance during walking. The investigators will record 3D coordinates of reflective markers placed on anatomical landmarks. These markers will be used to quantify changes in an individual's average peak lateral center of mass speed occurring each stride during treadmill walking.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
centimeters per second
  Pre-training assessment: number analyzed (Participants) | 18 | 17
  Pre-training assessment | 0.25 (0.14) | 0.22 (0.12)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 0.29 (0.13) | 0.23 (0.1)
  Post-training assessment: number analyzed (Participants) | 14 | 15
  Post-training assessment | 0.29 (0.15) | 0.27 (0.13)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 0.29 (0.12) | 0.24 (0.1)

19. Secondary Outcome: Step Width
Description: The investigators will perform biomechanical laboratory assessments to make quantitative measures of changes in dynamic balance during walking. The investigators will record 3D coordinates of reflective markers placed on anatomical landmarks. These markers will be used to quantify changes in an individual's preferred step width (lateral distance between calcaneal markers) during treadmill walking.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
meters
  Pre-training assessment: number analyzed (Participants) | 18 | 17
  Pre-training assessment | 0.27 (0.05) | 0.26 (0.06)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 0.26 (0.04) | 0.24 (0.06)
  Post-training assessment: number analyzed (Participants) | 14 | 15
  Post-training assessment | 0.26 (0.04) | 0.25 (0.06)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 0.26 (0.04) | 0.26 (0.06)

20. Secondary Outcome: Step Length
Description: The investigators will perform biomechanical laboratory assessments to make quantitative measures of changes in dynamic balance during walking. The investigators will record 3D coordinates of reflective markers placed on anatomical landmarks. These markers will be used to quantify changes in an individual's preferred step length (anterior - posterior distance between calcaneal markers) during treadmill walking.
Time Frame: as for outcome 1
Population: A total of 36 participants were analyzed
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treadmill Group | Movement Amplification Group
Number analyzed (Participants) | 18 | 18
meters
  Pre-training assessment: number analyzed (Participants) | 18 | 17
  Pre-training assessment | 0.27 (0.12) | 0.28 (0.16)
  Mid-training assessment: number analyzed (Participants) | 14 | 16
  Mid-training assessment | 0.37 (0.15) | 0.41 (0.11)
  Post-training assessment: number analyzed (Participants) | 14 | 16
  Post-training assessment | 0.41 (0.17) | 0.45 (0.13)
  Follow-up assessment: number analyzed (Participants) | 14 | 14
  Follow-up assessment | 0.39 (0.15) | 0.43 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored for each participant for an average of 6 months.
Arm/Group | Treadmill Group | Movement Amplification Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 3/18 | 3/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treadmill Group (N=18) | Movement Amplification Group (N=18)
Cardiovascular Issues (Cardiac disorders) | 1 (1) | 1 (1) — Blood Pressure medication
Musculoskeletal Injury / Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — Pain in lower limbs or back

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT04340063/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT04340063/ICF_000.pdf